CLINICAL TRIAL: NCT00191997
Title: Optimal Treatment Duration With Olanzapine Following Remission of Manic or Mixed Episode. An Open-Label, Randomized Trial Comparing Two Treatment Strategies.
Brief Title: Optimal Length of Treatment Continuation With Olanzapine After Remission of Manic or Mixed Episode
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8834; F1D-XM-HGLW
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2006-07-25 (Estimated); Status verified 2006-07

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Olanzapine

INTERVENTIONS:
Drug: Olanzapine

SUMMARY:
This is a randomized, parallel, open-label study of patients who have responded to treatment in the acute phase of their manic or mixed episode, with or without psychotic symptoms, with olanzapine in mono or co-therapy, and who are in syndromic and symptomatic remission at the time of enrollment into the study.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients, male or female, at least 18 years old
* Patient or legal representative must understand the study and sign an informed consent document before any study procedure
* Must have a diagnosis of Bipolar Disorder type I and have a recent manic or mixed episode, with or without hospitalization, according to DSM-IV-TR criteria.
* Patients must be in syndromic and symptomatic remission, following DSM-IV-IR criteria, for the manic or mixed episode, at the time of study entry, with a total score for YMRS less than or equal to 12 and total store for HAMD less than or equal to 8 at visit 1 and 2.
* Remission must have been achieved taking olanzapine in mono or co-therapy, and it must have been maintained until study entry.
* Patients must have had, at least, 2 manic or mixed episodes within 3 years of the study entry, taking into account the current one.

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry, or with a study drug in other clinical trial
* Patients without symptoms or manic or mixed episode within one month of study entry.
* Confirmed diagnoses of Schizophrenia or other psychotic disorders (schizophreniform disorder, schizoaffective disorder, delusional disorder, brief psychotic disorder, shared psychotic disorder, substance-induced or medical condition psychotic disorder, psychotic disorder NOS),following DSM-IV-TR criteria.
* Patients that have achieved remission with ECT (electro convulsive therapy) in addition to psychopharmacological treatment
* Drug dependence or abuse, if it is a primary diagnose and the mood disorder is due to his administration
* Patients that at the time of study entry or at any other time of study, need treatment with antiepileptics or other substances with potential effect as mood stabilizers (i,e new antiepileptics different to Lithium, Valproic Acid and/or Carbamazepine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2004-10; Study Completion 2006-03

PRIMARY OUTCOMES:
The main objective of this study is to compare the efficacy in the prevention of relapse to manic, depressive, or
mixed episodes in two groups of bipolar I patients
who responded to open-label treatment with olanzapine in mono or co-therapy and who are in symptomatic and syndromic remission at the time of entering the study.
The first group will receive olanzapine for a period of
3 months following inclusion into the study; the second group will receive olanzapine for 12 months.
Relapses will be evaluated in terms of the total YMRS
(Young Mania Rating Scale) and HAMD-21 (the 21-item Hamilton Depression Rating Scale) scores.

SECONDARY OUTCOMES:
The secondary objectives posed by this study are the following:
To compare the efficacy of maintaining olanzapine for 3 months versus maintaining it for 12 months in
the improvement of symptomatology in patients who had achieved remission. To this end, the reductions
on the total YMRS score, YMRS specific non-psychotic
item scores, HAMD 21 total score, the scores on the
HAMD 21 specific mood-related items, the total and
positive scores on the BPRS (Brief Psychiatric Rating Scale), and the CGI BP S(Clinical Global Impression of Severity) with respect to baseline will be evaluated.
DSM IV TR criteria will be used for manic and
depressive episodes in order to assess syndromic improvement.
To compare the efficacy of long-term treatments by means of longitudinal assessment using the
general subscale of the CGI BP M (Clinical Global Impression - Modified) and proceeding to
intra- and intergroup analyses.
To evaluate the safety of maintenance treatment
with olanzapine and other coadjuvant medication
in both groups of follow up. To collect data
regarding treatment-derived adverse events,
changes in vital signs, laboratory analyses, and to measure the severity of possible extrapyramidal symptoms.
The Simpson Angus Scale, Barnes Akathisia Scale, and the Abnormal Involuntary Movement Scale (AIMS) will be used to assess the latter.
To determine the impact on resource utilization
the two treatment groups have. Direct costs derived
from hospital admissions, emergency room visits,
out-patient visits, home healthcare supports, as well as indirect costs derived from days out of work,
the patient's economic income, impact on the caregiver will also be quantified.
To assess the differences between groups
with respect to improvement in functioning and quality of life. The SF 36 Scale (the 36-Item Social Function Scale) will be applied.
To understand the degree of impact the illness provokes in relatives or caregivers
throughout the study. The self-report scale of
family burden (Escala de Carga Familiar - ECF) will be used for this purpose.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- Spain (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, León
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Lleida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Murcia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Ourense
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Salamanca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Tarrasa-Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Vitoria-Gasteiz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Zamora